CLINICAL TRIAL: NCT03859661
Title: A Study to Evaluate the Palatability of a Nutritional Support Biscuit (Fitabisc)
Acronym: Fitabisc
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was halted due to poor recruitment and date on the biscuits expiring
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SNE2445
Record Dates: First submitted 2017-01-24; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Fitabisc — Fitabisc is a chocolate cookie with vanilla cream filling which contains the most important antioxidants Vitamin C, Vitamin E, and the mineral Selenium. Fitabisc is not commercially available and for the purposes of this study it will be manufactured by Calerrific Ltd, which already produces a biscuit called CalBisc 100 as a simple calorie and nutritional supplement. Production takes place in a BRC Global Standard Grade A certified bakery operated by Farringford Foods in Portadown, Northern Ireland.

SUMMARY:
A study to evaluate the palatability of a nutritional support biscuit (Fitabisc) in patients about to undergo colorectal surgery.

DETAILED DESCRIPTION:
The question of preoperative supplementation raises another issue about how this might be provided for patients, especially at home.

The Chief Investigator has formulated a new biscuit 'Fitabisc' that contains the key antioxidants; vitamins C and E, selenium and glutamine. The advantage of a biscuit is that all ingredients of interest are combined within the one item and so this may be easier for patients to 'take' than other types of supplement. A survey involving 17 community pharmacies in England and Northern Ireland found that 60% of patients aged 60 - 89 years had difficulty swallowing tablets and capsules. The consistency of the biscuit is softer than traditional shortbread and crumbs readily which we hope will make it easy to eat.

The aim of this study is to test the palatability of Fitabisc and whether patients undergoing abdominal surgery can eat it in the desired quantities for 10 days before they are admitted to hospital.

In summary, most studies to date have looked perioperative or postoperative supplementation with antioxidants alone. No attempt has been made to do this using a palatable biscuit that would facilitate preoperative oral supplementation. If this study confirms the palatability of the biscuit and there is adherence to eating it then it would be our intention to set up a prospective randomized study in which the potential efficacy of Fitabisc would be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 16 and 80 years inclusive.
* Patients who are having colorectal surgery.
* Patients who are able to give voluntary, written informed consent to participate in the study and from whom written consent has been obtained.

Exclusion Criteria:

* Those who cannot or do not provide informed consent
* Patients with a known or suspected allergy to any of the ingredients of Fitabisc e.g. gluten or dairy products
* Patients with one of the following co-morbidities:

  * Haemochromatosis
  * Thalassaemia
  * Kidney disease
  * Liver disease
  * Reye syndrome
* Patients who already take supplements of vitamin C, E, selenium or glutamine.
* Patients with type 1 diabetes, or type 2 diabetes that requires them to have insulin or a hypoglycaemic drug such as Metformin.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-12; Primary Completion 2017-09-11 (Actual); Study Completion 2017-09-11 (Actual)

PRIMARY OUTCOMES:
Adherence to dose | 10 days
  Patients to keep a diary of their consumption
Palatability of biscuit | 10 days
  Study will measure palatability on a standard Likert scale after 10 days

SECONDARY OUTCOMES:
Progress of patients following surgery | 4-6 weeks post op.
  Adverse event collection - via patient reported outcomes and review of patient notes following surgery
Collection of events that might be associated with the ingredients of the biscuit. | 4-6 weeks post op.
  Adverse event collection - via patient reported outcomes and review of patient notes following surgery

CONTACTS AND LOCATIONS:
Overall Officials: John Macfie, MBChB, MD, Principal Investigator — York Teaching Hospital NHS Foundation Trust
Locations (1):
- York Teaching Hospital NHS Foundation Trust, York, United Kingdom